CLINICAL TRIAL: NCT04372485
Title: Leveraging Health Information Technology to Reduce Health Disparities in Adolescent Health Outcomes: A Patient-Centered Approach
Brief Title: Using Mobile Health (mHealth) to Improve STI Treatment Adherence Among Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Monika Goyal, Associate Professor of Pediatrics and Emergency Medicine, Children's National Research Institute
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro0001427
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Sexually Transmitted Diseases
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth (Other): Adolescents enrolled in this arm will receive treatment-related text messages.
  Interventions: Behavioral: mHealth Intervention
- Usual care (No Intervention): Adolescents in this arm will receive usual care.

INTERVENTIONS:
Behavioral: mHealth Intervention — Adolescents will receive text messages to facilitate treatment adherence
  Arms: mHealth

SUMMARY:
We will conduct a randomized trial to compare differences in sexually transmitted infection (STI) treatment adherence between patients receiving text messages versus those receiving usual care (e.g. no text messages). We hypothesize that STI treatment adherence will be 20% higher among patients randomized to receipt of two-way text messaging services.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent patients seen in the Emergency Department who test positive for gonorrhea, chlamydia, or pelvic inflammatory disease and are prescribed outpatient antibiotic treatment.

Exclusion Criteria:

* Patients will be excluded if they are unable to understand English, are critically ill, have cognitive impairment or if they do not have access to a cellular telephone with text messaging capabilities.

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
STI treatment adherence | 1-21 days after prescription filling
  Proportion of study participants who complete their medication as prescribed by self-report

SECONDARY OUTCOMES:
STI treatment receipt | 1-21 days after STI diagnosis
  Proportion of study participants who receive STI treatment; measured by prescription filling and/or receiving treatment at a healthcare facility

CONTACTS AND LOCATIONS:
Overall Officials: Monika Goyal, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No